CLINICAL TRIAL: NCT04551573
Title: A Study of the Pharmacokinetic and Pharmacodynamic Interactions Between Bictegravir, Tenofovir Alafenamide and Rifapentine in Healthy Adult Subjects
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000027436
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Tuberculosis; Hiv
Keywords: Pharmacokinetic and Pharmacodynamic Interactions
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rifapentine daily (Experimental): In addition to taking Biktarvy for four weeks, participants will also take Rifapentine dosed daily for four weeks (10mg/kg; 600 mg dose)
  Interventions: Drug: Rifapentine daily
- Rifapentine weekly (Experimental): In addition to taking Biktarvy for four weeks, participants will also take Rifapentine dosed weekly for another four more weeks (15 mg/kg; 900mg dose)
  Interventions: Drug: Rifapentine weekly

INTERVENTIONS:
Drug: Rifapentine daily — In addition to taking Biktarvy for four weeks, participants will also take Rifapentine dosed daily for four weeks (10mg/kg; 600 mg dose)
  Arms: Rifapentine daily
Drug: Rifapentine weekly — In addition to taking Biktarvy for four weeks, participants will also take Rifapentine dosed weekly for another four more weeks (15 mg/kg; 900mg dose)
  Arms: Rifapentine weekly

SUMMARY:
This is a single-center, open-label, fixed sequence, pharmacokinetic interaction study between bictegravir and tenofovir alafenamide with rifapentine dosed either daily or weekly.

Primary Aims

* To assess the effect of once-weekly rifapentine on the steady-state PK of BIC
* To assess the effect of once-daily rifapentine on the steady-state PK of BIC

Secondary Aims

* To assess the effect of daily dosed rifapentine on steady-state PK of TAF (measured as plasma and IC concentrations of TFV-DP)
* To assess the effect and timing of interactions of weekly dosed rifapentine on steady-state PK of TAF (measured as plasma and IC concentrations of TFV-DP)
* To assess the safety of BIC/TAF/FTC when coadministered with once-weekly or once-daily rifapentine

DETAILED DESCRIPTION:
Subjects will receive once-daily Biktarvy for 4 weeks to ensure all moieties of interest reach steady-state prior to the baseline PK assessment. Thereafter, subjects will be enrolled in one of two groups for PK analysis as follows:

Group one will continue Biktarvy and have rifapentine dosed daily for 4 weeks (10 mg/kg; 600mg dose).

Group two will continue Biktarvy and have rifapentine dosed weekly for 4 weeks (15 mg/kg; 900mg dose).

After 4 weeks of Biktarvy dosing, subjects will have a baseline intensive PK of plasma bictegravir (BIC), tenofovir alafenamide (TAF), tenofovir (TFV) levels at all time points, and peripheral blood mononuclear cells (PBMCs) will be collected at 24 hours post-dose for IC TFV-DP. This will occur prior to receiving their first dose of directly observed oral rifapentine co-administered with Biktarvy, thus serving as their own control. Rifapentine will thereafter be administered by directly observed therapy (DOT) or ingestion monitored by smart phone application (e.g., Time Stamp App or other phone app platform). Intensive PK assessments will be repeated after 4 weeks of RPT dosing for both Group 1 and 2.

Intensive PK sampling will be performed at time 0 (pre-dose), 15 and 30 min; 1, 2, 3, 4, 8, 12 and 24 hours post-dose with BIC/TAF/FTC alone and when coadministered with rifapentine. Plasma will be isolated at all time points, and PBMCs will be isolated at 24 hours post-dose.

PK levels will be measured by colleagues at the Colorado Antiviral Pharmacology (CAVP) Laboratory at the University of Colorado Anschutz Medical Campus. Plasma concentrations of BIC, TAF, TFV, and IC TFV-DP in PBMCs will be measured by liquid chromatography-tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults deemed by the investigator to have acceptable medical history, physical examination, 12 lead electrocardiogram, and clinical laboratory evaluations
* Body weight > or equal to 50 kg for males and females
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive. BMI = weight (kg)/ height (m2)
* Male or females, ages > or equal to 18 years

Exclusion Criteria:

* Positive screening HIV+ as determined by standard serologic and molecular assays or suspected acute HIV infection in the opinion of the clinician
* Subjects with AST, ALT or bilirubin > 2.5X the upper limit of normal.
* Hemoglobin < 9 g/dL, and platelet count < 75, 000/mm3.
* Positive serum or urine for HCG.
* Positive or indeterminate interferon gamma release assay
* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* Proven or suspected acute hepatitis at the time of study entry
* Untreated and /or active Hepatitis B or C infection or chronic liver disease with liver cirrhosis (as determined by biopsy or non-invasive testing)
* Current or recent (within 3 months) gastrointestinal disease that would interfere with the conduct or interpretation of the study.
* Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Evidence of organ dysfunction or any clinically relevant deviations (as determined by the investigator) from the norms observed in the general population regarding physical examination, vital signs, ECG or clinical laboratory determinations.
* Any major surgery within 4 weeks of enrollment. Minor surgical procedures requiring local anesthesia are exceptions.
* Signs and symptoms of or known pulmonary or extra-pulmonary tuberculosis
* A history of porphyria
* History of or known allergy to rifamycins.
* Exposure to any investigational drug within 4 weeks of enrollment and throughout the study.
* Use of any agent, within 2 weeks of dosing, that is known to induce or inhibit drug metabolizing enzymes (e.g., cimetidine and compounds in the barbiturate and phenothiazine classes), affect renal tubular secretion (e.g., probenecid, beta-lactam antibiotics), gastrointestinal motility (e.g., metoclopramide, propantheline, loperamide, or narcotic analgesics or opioids other than methadone), or uric acid metabolism (e.g., allopurinol) or gastrointestinal pH (including antacids, H2-receptor antagonists, proton pump inhibitors etc.).
* Use of any prescription drugs (other than methadone) or over-the-counter acid controllers within 2 weeks prior to enrollment and throughout the study.
* Positive breathalyzer alcohol test, or positive urine screen for barbiturates, benzodiazepines, amphetamines, THC, cocaine or opioids other than methadone at screening.
* Use of any other drugs, including over-the-counter medications (e.g., acetaminophen) and herbal preparations, within 1 week prior to enrollment and throughout the study. Use of any other concurrent medication, must be discussed with the medical monitor prior to use.
* Use of an oral, injectable or implantable hormonal contraceptive agent within 3 months of enrollment and throughout the study.
* History of any significant drug allergy, drug rash or sensitivity to any class of drugs relevant to the study drugs.
* Use of St. John's Wort (Hypericum) within four weeks prior to study enrollment and throughout the study.
* Consumption of grapefruit or grapefruit juice within 1 week of study entry and throughout the study.
* Women who are pregnant or breastfeeding
* Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks before and after the study.
* WOCBP using a prohibited contraceptive method (oral, injectable or implantable hormonal agents)
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on screening, enrollment or prior to study drug administration.
* Donation of blood or plasma to a blood bank or as part of a clinical study (except at screening visit) within 4 weeks of enrollment.
* Blood transfusion within 4 weeks of enrollment.
* Inability to tolerate oral medications.
* Inability to tolerate venipuncture and/or absence of secure venous access.
* Inability to refrain from smoking during in-residence period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Plasma area under the curve (AUC) of Bictegravir between groups | 8 weeks
  Determining plasma AUCtau of Bictegravir when co-administered with rifapentine as once-daily or once-weekly
Maximum plasma concentrations(Cmax) of Bictegravir between groups | 8 weeks
  Determining Cmax of Bictegravir when co-administered with rifapentine as once-daily or once-weekly
Concentrations at the end of dosing interval (Ctau) of Bictegravir between groups | 8 weeks
  Determining Ctau of Bictegravir when co-administered with rifapentine as once-daily or once-weekly
Time to total maximum plasma concentrations (Tmax) of Bictegravir between groups | 8 weeks
  Determining Tmax of Bictegravir when co-administered with rifapentine as once-daily or once-weekly

SECONDARY OUTCOMES:
Plasma area under the curve (AUC) of tenofovir alafenamide (TAF) between groups | 8 weeks
  Determining plasma AUCtau of TAF when co-administered with rifapentine as once-daily or once-weekly
Maximum plasma concentrations(Cmax) of TAF between groups | 8 weeks
  Determining Cmax of TAF when co-administered with rifapentine as once-daily or once-weekly
Steady-state Intracellular (IC) concentration changes of tenofovir-diphosphate (TFV-DP) | 8 weeks
  Determining steady-state intracellular (IC) concentration changes of TFV-DP when co-administered with rifapentine at two different dosing intervals (daily and weekly)
Adverse Events of medications | 8 weeks
  Adverse events of co-administration of rifapentine with BIC/TAF/ Emtrictabine (FTC)

CONTACTS AND LOCATIONS:
Overall Officials: Onyema Ogbuagu, MBBCh, FACP, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes